CLINICAL TRIAL: NCT03607240
Title: The Effect of Ultrasound-guided Alveolar Recruitment on Postoperative Atelectasis in Patients Receiving Laparoscopic Gynecological Surgery
Brief Title: Ultrasound-guided Alveolar Recruitment in Laparoscopic Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-1805-148-948
Record Dates: First submitted 2018-07-01; First posted 2018-07-31 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Pulmonary Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LUS-guided alveolar recruitment (Experimental): Lung ultrasound-guided alveolar recruitment maneuver will be performed
  Interventions: Procedure: lung ultrasound-guided alveolar recruitment
- conventional alveolar recruitment (Active Comparator): Alveolar recruitment maneuver will be provided with positive pressure of 30 cmH2O for 10 seconds.
  Interventions: Procedure: conventional alveolar recruitment

INTERVENTIONS:
Procedure: lung ultrasound-guided alveolar recruitment — Alveolar recruitment maneuver will be performed under lung ultrasound-guidance. Positive pressure will be not exceed 40cmH2O and duration of positive pressure inflation will not exceed 10 seconds.
  Arms: LUS-guided alveolar recruitment
Procedure: conventional alveolar recruitment — Alveolar recruitment will be provided with positive pressure of 30cmH2O for 10 seconds
  Arms: conventional alveolar recruitment

SUMMARY:
The study aims to compare the degree of atelectasis between ultrasound-guided alveolar recruitment group and conventional alveolar recruitment group in patients receiving laparoscopic gynecologic surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled to undergo elective laparoscopic gynecological surgery (laparoscopic ovarian cystectomy or laparoscopic salpingo-oophorectomy or laparoscopic hysterectomy or laparoscopic myomectomy) under general anesthesia, with ASA physical status classification I or II

Exclusion Criteria:

* Previous history of lung surgery
* Patients having pneumonia, pneumothorax, or pleural effusion in preoperative chest X-ray
* Patients with COPD, emphysema
* Patients with previous history of pneumothorax, or bullae
* Morbid cardiac disease
* Adolescent aged < 18 years
* Anticipated duration of surgery < 1 hour

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
modified lung ultrasound score at the end of surgery | At the end of surgery
  Both lung ultrasound scores can be calculated by adding up the 12 individual pulmonary quadrant scores yielding a score between 0 (no aeration loss) and 36 (complete aeration loss).

SECONDARY OUTCOMES:
modified lung ultrasound score at post-anesthesia care unit (PACU) | intraoperative
  Both lung ultrasound scores can be calculated by adding up the 12 individual pulmonary quadrant scores yielding a score between 0 (no aeration loss) and 36 (complete aeration loss).
incidence of atelectasis diagnosed by ultrasonography | intraoperative
  the presence of atelectasis by ultrasonography
arterial blood gas analyses | intraoperative
  PaO2, PaCO2, SaO2, O2 index (PaO2/FiO2)
incidence of postoperative complications | during the postoperative period until discharge from hospital, an average of 3 days
  fever, pneumonia, atelectasis diagnosed by chest X-ray
intraoperative mean arterial pressure | intraoperative
  mean arterial pressure in mmHg
intraoperative SpO2 | intraoperative
  SpO2 in %
intraoperative peak airway pressure | intraoperative
  peak airway pressure in cmH2O
Incidence of postoperative shoulder pain at POD #1 | assessed at postoperative day 1
  patients will be asked whether they have shoulder pain or not, using NRS (0 to 10) scale

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Jin-Tae Kim, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monastesse A, Girard F, Massicotte N, Chartrand-Lefebvre C, Girard M. Lung Ultrasonography for the Assessment of Perioperative Atelectasis: A Pilot Feasibility Study. Anesth Analg. 2017 Feb;124(2):494-504. doi: 10.1213/ANE.0000000000001603. PMID 27669555
- [Background] Song IK, Kim EH, Lee JH, Ro S, Kim HS, Kim JT. Effects of an alveolar recruitment manoeuvre guided by lung ultrasound on anaesthesia-induced atelectasis in infants: a randomised, controlled trial. Anaesthesia. 2017 Feb;72(2):214-222. doi: 10.1111/anae.13713. Epub 2016 Nov 2. PMID 27804117
- [Derived] Park SK, Yang H, Yoo S, Kim WH, Lim YJ, Bahk JH, Kim JT. Ultrasound-guided versus conventional lung recruitment manoeuvres in laparoscopic gynaecological surgery: A randomised controlled trial. Eur J Anaesthesiol. 2021 Mar 1;38(3):275-284. doi: 10.1097/EJA.0000000000001435. PMID 33399385